CLINICAL TRIAL: NCT02268851
Title: A Multi-center Phase I/Ib Study Evaluating the Efficacy and Safety of the Novel PI3k Delta Inhibitor TGR-1202 in Combination With Ibrutinib in Patients With Select B-Cell Malignancies
Brief Title: A Phase I/Ib Safety and Efficacy Study of the PI3K-delta Inhibitor TGR-1202 and Ibrutinib in Patients With CLL or MCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: TG Therapeutics, Inc. (Industry); The Leukemia and Lymphoma Society (Other); Blood Cancer Research Partnership (Other)
Responsible Party: Principal Investigator, Matthew S. Davids, MD, Principal Investigators, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14-396; TGR-IB-105 (Other: TG Therapeutics)
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — umbralisib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLL (Experimental): Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  * Each Cycle = 28 days
  * TGR-1202 (oral): Starting on Day 1 administered daily.
  * Ibrutinib (oral): Starting on Day 1 administered daily.
  Interventions: Drug: TGR-1202; Drug: Ibrutinib
- MCL (Experimental): Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  * Each Cycle = 28 days
  * TGR-1202 (oral): Starting on Day 1 administered daily.
  * Ibrutinib (oral): Starting on Day 1 administered daily.
  Interventions: Drug: TGR-1202; Drug: Ibrutinib

INTERVENTIONS:
Drug: TGR-1202 — Capsules taken whole daily with water and with food
  Other Names: RP5264; Umbralisib
Drug: Ibrutinib — Capsules taken whole with water- Do not consume fish oil, vitamin E, grapefruit, or Seville oranges
  Other Names: Imbruvica; CRA-032765; PCI-32765

SUMMARY:
This research study will be evaluating the safety and efficacy of a study drug called TGR-1202 in combination with a known drug ibrutinib, also known as Imbruvica, as a possible treatment for Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) or Mantle Cell Lymphoma (MCL) that has come back or that has not responded to standard treatment.

DETAILED DESCRIPTION:
This research study is a Phase I and Ib combination clinical trial, which aims to both evaluate the safety of an investigational drug combination and also tries to define the appropriate dose of the investigational drug to evaluate in later clinical trials. "Investigational" means that the intervention is being studied. It also means that the FDA (U.S. Food and Drug Administration) has not approved TGR-1202 in the United States for use in MCL/CLL/SLL cancers.

TGR-1202 is a newly developed drug that may stop cancer cells from growing based on recent laboratory experiments. The results from these experiments suggest this drug may help to kill cancer cells when coupled with ibrutinib. In this research study, the safety and tolerability of TGR-1202 is being investigated to determine the highest dose that can safely be used in combination with ibrutinib. The study is also aimed to evaluate whether TGR-1202 has any effect on tumor growth (nodal response), and to determine the overall repsonse rate and duration of response in patients with CLL/SLL or MCL

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Mantle Cell Lymphoma (MCL), Chronic Lymphocytic Leukemia (CLL), or Small Lymphocytic Lymphoma (SLL)
* Adequate organ system function ( Absolute neutrophil count, Platelets,Bilirubin, Platelets, Aspartate transferase ,Alanine aminotransferase, Creatinine Clearance)
* Eastern Cooperative Group (ECOG) Performance status ≤ 2
* Ability to swallow and retain oral medication
* Female patients: must have negative serum pregnancy test at study screening/ all male partners must consent to use a medically acceptable method of contraception
* Willingness and ability to comply with trial and follow-up procedures, and give written informed consent

Exclusion Criteria:-

* Patients receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization) within 3 weeks of Cycle 1/Day 1,
* Autologous hematologic stem cell transplant within 3 months of study entry.
* Allogeneic hematologic stem cell transplant within 12 months.

  * Post-allo patients must not have active graft versus-host disease
* Evidence of active Hepatitis B,Hepatitis C or HIV infection.
* Active central nervous system involvement by lymphoma
* Requires treatment with strong CYP3A4/5 inhibitors
* Severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* QTcF >470 msec (QT interval, Fredericia calculation)
* Angina not well-controlled by medication
* Poorly controlled or clinically significant atherosclerotic vascular disease
* Presence of other active cancers, or history of treatment for invasive cancer within the past 2 years.
* Require warfarin for anticoagulation
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05 (Actual); Study Completion 2022-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davids, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Pacific Cancer Care, Monterey, California
  - St. Francis Hospital and Cancer Center, Hartford, Connecticut
  - Eastern Maine Medical Center/ Northern Light Cancer Care, Brewer, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davids MS, Kim HT, Nicotra A, Savell A, Francoeur K, Hellman JM, Bazemore J, Miskin HP, Sportelli P, Stampleman L, Maegawa R, Rueter J, Boruchov AM, Arnason JE, Jacobson CA, Jacobsen ED, Fisher DC, Brown JR; Blood Cancer Research Partnership of the Leukemia and Lymphoma Society. Umbralisib in combination with ibrutinib in patients with relapsed or refractory chronic lymphocytic leukaemia or mantle cell lymphoma: a multicentre phase 1-1b study. Lancet Haematol. 2019 Jan;6(1):e38-e47. doi: 10.1016/S2352-3026(18)30196-0. Epub 2018 Dec 14. PMID 30558987

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the Phase I portion of the study enrolled in outpatient clinic setting from 11/20/2014 to 12/22/2018 and to the Phase II study from 1/14/2016 to 5/29/2018. The MCL and CLL arms were enrolled independently of each other, and were allowed to begin enrolling to the protocol scheduled expansion independent of the other arm.
Groups:
- CLL: Phase I Cohort 1: Phase I Cohort 1 patients received oral agent TGR1202 400mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 420 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- MCL: Phase I Cohort 1: Phase I Cohort 1 patients received oral agent TGR1202 400mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 560 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- CLL: Phase I Cohort 2; MCL: Phase I Cohort 2: Phase I Cohort 2 patients received oral agent TGR1202 600mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 420 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- CLL: Phase I/II Cohort 3 (RPD2); MCL: Phase I/II Cohort 3 (RPD2): Phase I Cohort 3 patients received oral agent TGR1202 800mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 420 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
Period: Overall Study
Arm/Group | CLL: Phase I Cohort 1 | MCL: Phase I Cohort 1 | CLL: Phase I Cohort 2 | MCL: Phase I Cohort 2 | CLL: Phase I/II Cohort 3 (RPD2) | MCL: Phase I/II Cohort 3 (RPD2)
Started | 3 | 3 | 4 | 3 | 15 | 15
Completed | 2 | 0 | 3 | 0 | 8 | 4
Not Completed | 1 | 3 | 1 | 3 | 7 | 11
Not completed — Death | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Progressive Disease | 1 | 3 | 0 | 0 | 1 | 4
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Patient Compliance | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Co-Morbid Condition | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- MCL: Phase 1 Cohort 1: Phase I Cohort 1 patients received oral agent TGR1202 400mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 560 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- MCL: Phase I Cohort 2: Phase I Cohort 2 patients received oral agent TGR1202 600mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 560 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- CLL Phase I/IICohort 3 (RPD2): Phase I Cohort 3 patients received oral agent TGR1202 800mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 420 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- MCL Phase I/II Cohort 3 (RPD2): Phase I Cohort 3 patients received oral agent TGR1202 800mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 560 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- Total: Total of all reporting groups
Arm/Group | CLL: Phase I Cohort 1 | MCL: Phase 1 Cohort 1 | CLL: Phase I Cohort 2 | MCL: Phase I Cohort 2 | CLL Phase I/IICohort 3 (RPD2) | MCL Phase I/II Cohort 3 (RPD2) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 15 | 15 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 2 | 1 | 2 | 3 | 12
  >=65 years | 0 | 2 | 2 | 2 | 13 | 12 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 2 | 5 | 5 | 17
  Male | 1 | 3 | 1 | 1 | 10 | 10 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 3 | 4 | 2 | 15 | 15 | 41
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 3 | 15 | 15 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced a Dose Limiting Toxicity (DLT) During Phase I
Description: To assess the safety of TGR1202 in combination with ibrutinib relapsed or refractory CLL or MCL. DLT is based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. DLT refers to toxicities experienced at any time during the study treatment, defined as Grade 4 anemia; Grade 4 neutropenia lasting >7 days (while receiving growth factor support); Grade 4 thrombocytopenia lasting > 7 days; Grade ≥3 febrile neutropenia; and Grade ≥3 thrombocytopenia with Grade >2 hemorrhage;Grade ≥ 3 non-hematologic toxicity unresponsive to standard supportive care measure with the exception of asymptomatic Grade ≥3 lab abnormalities that resolve to ≤ Grade 1 or baseline within 7 days;treatment delay of ≥14 days due to unresolved toxicity; and non-hematologic toxicity of Grade 2 (at any time during treatment) that, in the judgment of the Investigators, Study Chair, and the Medical Monitor, is dose-limiting.
Time Frame: Participants were assessed every week or more often as needed during Cycle 1 or more often for up to 28 days to assess Dose-limiting toxicities (DLTs) during Phase I
Population: Patients who have been previously treated for MCL, CLL or SLL. MCL must have 1 measurable site of disease and have had received at least one prior standard therapy; CLL/SLL patients must have an indication for treatment according to 2008 ICWLL criteria and received at least one prior standard treatment regimen
Measure: Count of Participants; unit: Participants
Groups:
- MCL Phase I/II Cohort 3 (RPD2): Phase I Cohort 3 patients received oral agent TGR1202 800mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 420 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
Arm/Group | CLL: Phase I Cohort 1 | MCL: Phase 1 Cohort 1 | CLL: Phase I Cohort 2 | MCL: Phase I Cohort 2 | CLL Phase I/IICohort 3 (RPD2) | MCL Phase I/II Cohort 3 (RPD2)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 15 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on the 2008 IW-CLL criteria for CLL (Hallek et al., 2008) by Lugano Criteria ( Cheson et al,.24) for MCL.
Time Frame: At baseline, End of Cycle 2, End of Cycle 5, End of Cycle 9, End of Cycle 14 and approximately q6 months until C26, then investigator discretion thereafter
Population: all the patients were pooled together from ph1 and ph1b for the final efficacy analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CLL Cohort; MCL Cohort: Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  * Each Cycle = 28 days
  * TGR-1202 (oral): Starting on Day 1 administered daily.
  * Ibrutinib (oral): Starting on Day 1 administered daily.
Arm/Group | CLL Cohort | MCL Cohort
Number analyzed (Participants) | 21 | 21
percentage of participants | 95.2 [58.17 to 100] | 71.4 [39.98 to 100]

3. Secondary Outcome: Rate of Nodal Partial Response With Lymphocytosis (nPR)
Description: nPR will only be evaluated in CLL patients, defined as percentage of patients achieved nodal PR. As per Cheson et al., 2012, patients who achieve a radiographic PR but continue to have a lymphocytosis with >5,000 B-lymphocytes per μL are considered to have a nodular partial response, also known as PR with lymphocytosis, due to the fact that they appear to derive a similar clinical benefit from BCR inhibitors as patients who achieve a traditional PR.
Time Frame: as for outcome 2
Population: all the patients were pooled together from ph1 and ph1b for the final efficacy analysis
Measure: Number; unit: percentage of patients
Arm/Group | CLL Cohort
Number analyzed (Participants) | 21
percentage of patients | 71.4

4. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last dsease assessment.
Time Frame: Disease will be evaluated at baseline, cycle 1 day 1,8,15,22 and cycle 2 day 1,15, and cycle 3-6 on day1, and every 2 cycles until cycle 12, then every 3 cycles thereafter. In long-term follow-up, survival will be followed every 3 cycles up to 2 years.
Population: all the patients were pooled together from ph1 and ph1b for the final efficacy analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CLL Cohort | MCL Cohort
Number analyzed (Participants) | 21 | 21
months | 82.66 [55.23 to NA] — Upper limit not statistically reachable using KM | 26.87 [10.09 to NA] — Upper limit not statistically reachable using KM

5. Secondary Outcome: Median Duration of Overall Response (DOR)
Description: Duration of Overall Response (DOR), estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per 2008 IWCLL Criteria, until the first date that recurrent or progressive disease is objectively documented. Patients without progressive disease are censored at the date of last disease assessment.
Time Frame: Disease response will be evaluated at baseline, cycle 1 day 1,8,15,22 and cycle 2 day 1,15, and cycle 3-6 on day1, and every 2 cycles until cycle 12, then every 3 cycles thereafter.
Population: all the patients were pooled together from ph1 and ph1b for the final efficacy analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CLL Cohort | MCL Cohort
Number analyzed (Participants) | 21 | 21
months | 80.36 [46.42 to NA] — Upper limit not statistically reachable using KM | 42.32 [9.17 to NA] — Upper limit not statistically reachable using KM

ADVERSE EVENTS:
Time Frame: Adverse events are assessed at minimum every week during cycle 1, on days 1 and 15 of cycle 2, every Day 1 of cycles 3-6 where every cycle is 28 days. Cycles 8-12, participants are evaluated every other cycle on Day 1, and then every 3 cycles Cycle 12 onward to Cycle 36, then every 6 cycles on Day 1 thereafter. The DLT period was the first 28 days of treatment during Phase I. AEs were assessed up to 30 days after drug discontinuation.
Description: Maximum grade toxicity by type-Serious AEs were defined as per DFCI criteria: Any grade 2 or 3 unexpected and treatment related event, unexpected grade 4 events, all grade 5 events regardless of attribution to study treatment. Includes events deemed medically important by overall PI. Other AEs were defined as events with the attribution of at least possibly related to the study treatment that did not meet the SAE criteria. CTCAE 4.0 was used in investigator assessment and lab value review.
Groups:
- CLL: Phase I/IICohort 3 (RPD2); MCL: Phase I/II Cohort 3 (RPD2): Phase I Cohort 3 patients received oral agent TGR1202 800mg daily on days 1-28 of a 28 day cycle and ibrutinib orally 420 mg daily on days 1-28 of a 28 day cycle. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
Arm/Group | CLL: Phase I Cohort 1 | MCL: Phase I Cohort 1 | CLL: Phase I Cohort 2 | MCL: Phase I Cohort 2 | CLL: Phase I/IICohort 3 (RPD2) | MCL: Phase I/II Cohort 3 (RPD2)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/4 | 1/3 | 2/15 | 3/15
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 0/4 | 1/3 | 3/15 | 5/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 15/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLL: Phase I Cohort 1 (N=3) | MCL: Phase I Cohort 1 (N=3) | CLL: Phase I Cohort 2 (N=4) | MCL: Phase I Cohort 2 (N=3) | CLL: Phase I/IICohort 3 (RPD2) (N=15) | MCL: Phase I/II Cohort 3 (RPD2) (N=15)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Suspected adrenal insufficiency and suspected disease progression- both without autopsy
Paraspinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLL: Phase I Cohort 1 (N=3) | MCL: Phase I Cohort 1 (N=3) | CLL: Phase I Cohort 2 (N=4) | MCL: Phase I Cohort 2 (N=3) | CLL: Phase I/IICohort 3 (RPD2) (N=15) | MCL: Phase I/II Cohort 3 (RPD2) (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 3
Alkaline phosphatase increased (Investigations) | 2 | 1 | 3 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 3 | 2 | 15 | 7
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 4 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 3 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 1 | 2 | 7 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1 | 5 | 3
Bloating (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 1 | 3 | 4
Blurred vision (Eye disorders) | 1 | 0 | 1 | 1 | 3 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 9 | 7
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 7 | 3
Creatinine increased (Investigations) | 1 | 1 | 1 | 1 | 5 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 2 | 3 | 10 | 12
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 2 | 6 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 5 | 4
Edema limbs (General disorders) | 2 | 0 | 2 | 1 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 2
Fatigue (General disorders) | 3 | 2 | 3 | 3 | 12 | 13
Fever (General disorders) | 1 | 1 | 1 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 2 | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 2
Headache (Nervous system disorders) | 2 | 2 | 2 | 1 | 4 | 6
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 2 | 1
Hematoma (Vascular disorders) | 1 | 1 | 1 | 0 | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 3 | 14 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 1 | 3 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 3
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1 | 3 | 5
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 3 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 3 | 4 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2 | 7 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 6 | 4
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 3 | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2 | 6
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 3 | 5 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 3 | 6
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 1 | 3 | 4
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 5 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
Localized edema (General disorders) | 2 | 0 | 1 | 1 | 1 | 3
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 5 | 4
Lymphocyte count decreased (Investigations) | 0 | 1 | 2 | 1 | 1 | 6
Lymphocyte count increased (Investigations) | 3 | 2 | 2 | 0 | 11 | 2
Malaise (General disorders) | 0 | 0 | 0 | 1 | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 4 | 2
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 3 | 3
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 8 | 9
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 3 | 2 | 0 | 13 | 7
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1 | 2 | 2
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Platelet count decreased (Investigations) | 2 | 3 | 2 | 2 | 15 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 6 | 3
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0
Skin infection (Infections and infestations) | 1 | 0 | 2 | 0 | 2 | 2
Skin/subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 — Various types of non specific rashes
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 3 | 1 | 0 | 0 | 6 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2 | 5
Weight gain (Investigations) | 0 | 0 | 0 | 1 | 4 | 2
Weight loss (Investigations) | 0 | 1 | 2 | 0 | 0 | 2
White blood cell decreased (Investigations) | 2 | 2 | 2 | 0 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02268851/Prot_SAP_000.pdf